CLINICAL TRIAL: NCT05614128
Title: Validation of Cutaneous Nerve Demyelination in Diagnosis and Treatment of CIDP
Status: Terminated | Type: Observational
Why Stopped: Difficulty with Recruitment, Lack of Funding
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Principal Investigator, Amanda Peltier, Professor, Vanderbilt University Medical Center
Other Study IDs: VR64081
Record Dates: First submitted 2022-10-31; First posted 2022-11-14 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: CIDP
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 2 mm punch skin biopsies will be obtained at the index finger on the palm side of the non-dominant hand.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: IVIg — Patients will be treated with IVIg as recommended by expert guidelines for treatment of CIDP under care of their primary neurologist. This will not be provided by the study.

SUMMARY:
The goal of this observational study is to learn about chronic inflammatory demyelinating polyneuropathy. The main question the investigators would like to answer is 1) can skin biopsy identify demyelination better than nerve conduction studies (electrical tests of the nerves)? and 2) how do nerves improve after treatment in CIDP? Participants will be asked to undergo skin biopsy of the finger at baseline and at 3 months and 6 months after treatment with IVIG (which is the FDA approved treatment for CIDP).

DETAILED DESCRIPTION:
Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP) is an autoimmune disorder that can cause severe weakness and numbness, difficulty walking if untreated. CIDP is a disorder where the myelin or outside covering of the nerves which protect nerves and speed conduction are damaged by the immune system. The typical way CIDP is diagnosed is by performing electrical stimulation of the nerves (nerve conduction study or NCS) which may not be very accurate in identifying CIDP. The investigators also are not clear on how CIDP nerve impairment improves with treatment after IVIg, which is the recommended treatment. This study uses skin biopsy of the finger to look at the nerves and see if abnormalities of myelin such as segmental demyelination (loss of myelin along the course of the nerve) can be detected under microscope. The investigators will repeat the skin biopsy during treatment with IVIg (brand Privigen which is FDA approved for CIDP) to determine how IVIg improves nerves during treatment. The investigators hope this study will provide both better ways to diagnose patients with CIDP as well as inform doctors on how CIDP can improve with treatment.

The investigators are recruiting patients newly diagnosed or within 6 months of diagnosis to study the use of skin biopsies in diagnosis of CIDP. The investigators are also repeating skin biopsies at 3 months and 6 months to measure improvement in nerve demyelination.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥ 18 years) with definite or probable CIDP according to the EFNS/PNS criteria may enter the trial within 12 months of treatment onset or treatment naïve patients. Written informed consent is obtained by the local investigator before entry into the study.

  2. IVIg treatment of 0.8 up to 1.2 g/kg per 30 days will be allowed up to 6 months. It is expected some patients may be on variable treatment regimens, and as along as they are not significantly declining, efforts will be made to continue treatment regimens already instituted.

  3. Prednisone in doses up to 20 mg /day will be allowed as long as dose has been stable for 90 days and is not being escalated or tapered during study.

  4. Previous plasma exchange will be allowed as long as it is not continued during the study.

Exclusion Criteria:

* 1. Other causes of polyneuropathy, multifocal motor neuropathy, diabetes mellitus, alcohol, family history of neuropathy, monoclonal gammopathy or malignancy, history of drug or toxin exposure, which could reasonably cause neuropathy. Coexistent monoclonal gammopathy will also be used as an exclusion as these patients may not have the same response to IVIg.

  2. Any other disease that may cause neurological symptoms and signs or that may interfere with treatment or outcome assessments.

  3. Severe conditions that may interfere with an evaluation of the study product or satisfactory conduct of the study such as current malignancy or history of allogeneic bone marrow/stem cell transplant, cardiac insufficiency (New York Heart Association Classes III/IV), cardiomyopathy, cardiac arrhythmia requiring treatment, unstable or advanced ischemic heart disease, congestive heart failure or severe hypertension, chronic kidney disease deemed too severe to safely use IVIg, known hyperprolinemia, known bleeding disorders, severe skin disease at the planned injection sites or biopsy site, alcohol, drug or medication abuse.

  4. History of keloids or other reactions to local anesthetic making skin biopsies unsafe.

  5. Patients with the following laboratory results:
  1. Positive result at screening on any of the following viral markers: human immunodeficiency virus-1 or 2, or hepatitis B or C virus.
  2. Abnormal laboratory parameters: creatinine greater than 1.5 times the upper limit of normal (ULN), blood urea nitrogen greater than three times the ULN if the increase is related to potential kidney disease, or hemoglobin less than 10 g/dL

  b. Abnormal laboratory parameters: creatinine greater than 1.5 times the upper limit of normal (ULN), blood urea nitrogen greater than three times the ULN if the increase is related to potential kidney disease, or hemoglobin less than 10 g/dL 6. Fulfilling the following general criteria: inability to comply with study procedures and treatment regimen; mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the study; pregnancy or nursing mother; intention to become pregnant during the course of the study; female patients of childbearing potential either not using or not willing to use a medically reliable method of contraception for the entire duration of the study or not sexually abstinent for the entire duration of the study or not surgically sterile; participation in another clinical study or use of another investigational medicinal product within the same time period of the study.

  7. Additional medications and treatments other than prednisone and IVIg for treatment of CIDP such as azathioprine, mycophenolate, rituximab and ongoing plasma exchange as this will either confound or interfere with effects of IVIg.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed patients with CIDP prior or within 12 months of treatment with IVIg.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-09-19 (Actual)

PRIMARY OUTCOMES:
Percentage of cutaneous nerves with segmental demyelination | 6 months
  Number of nerve fibers with demyelination visualized under microscopy will be calculated per biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Wende Fedder, Rn, Study Director — Vanderbilt University Medical Center; Diana Davis, RN, Study Director — Vanderbilt University Medical Center
Locations (1):
- Peltier Amanda, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-10-04): https://cdn.clinicaltrials.gov/large-docs/28/NCT05614128/Prot_ICF_000.pdf